CLINICAL TRIAL: NCT01091090
Title: Cognitive Behavioral Smoking Cessation Intervention for Adults With Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: W. Michael Hooten, MD, Mayo Clinic Foundation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09-006264
Record Dates: First submitted 2010-03-10; First posted 2010-03-23 (Estimated); Last update posted 2012-05-25 (Estimated); Status verified 2012-05

CONDITIONS: Smoking Cessation
Keywords: Smoking cessation; Nicotine dependence; Chronic pain
MeSH Terms: conditions — Smoking Cessation; Tobacco Use Disorder; Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive behavioral (Experimental): Subjects with receive a cognitive behavioral intervention for smoking cessation
  Interventions: Behavioral: Cognitive behavioral
- Control (Active Comparator): Treatment as usual
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Cognitive behavioral — Cognitive behavioral intervention for smoking cessation
  Other Names: Cognitive; Behavioral; Smoking Cessation
  Arms: Cognitive behavioral
Behavioral: Control — Treatment as usual
  Arms: Control

SUMMARY:
Millions of individuals with chronic pain smoke and our preliminary research suggests that currently available strategies to help people quit smoking may not be effective for individuals with chronic pain. This is important in that smokers with chronic pain have worse pain-related health outcomes compared to nonsmokers with chronic pain. The primary aim of this research project is to develop a smoking cessation intervention for specific use in an outpatient clinical setting for smokers with chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* Chronic pain
* Age > 18 years
* Cigarette smoker > 10 per day

Exclusion Criteria:

* Concurrent substance use disorder other than nicotine dependence
* Concurrent major psychiatric disorder

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2009-11; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
The key measurement to be used to assess the effect of the experimental intervention will be the status of cigarette smoking at 6-month follow-up. | 6 months
  The smoking status will be determined by assessing the 7-day point prevalence use of cigarettes which is defined as the use of any cigarettes within the preceding 7 days of the follow-up date at 6-months.

SECONDARY OUTCOMES:
A key secondary outcome measure will be self-report pain severity at 6-months following completion of the experimental intervention. | 6 month

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Pain Rehabilitation Center, Rochester, Minnesota, United States

REFERENCES:
- [Background] Hooten WM, Townsend CO, Bruce BK, Shi Y, Warner DO. Sex differences in characteristics of smokers with chronic pain undergoing multidisciplinary pain rehabilitation. Pain Med. 2009 Nov;10(8):1416-25. doi: 10.1111/j.1526-4637.2009.00702.x. Epub 2009 Sep 1. PMID 19732372
- [Background] Hooten WM, Townsend CO, Bruce BK, Warner DO. The effects of smoking status on opioid tapering among patients with chronic pain. Anesth Analg. 2009 Jan;108(1):308-15. doi: 10.1213/ane.0b013e31818c7b99. PMID 19095867
- [Background] Hooten WM, Townsend CO, Bruce BK, Schmidt JE, Kerkvliet JL, Patten CA, Warner DO. Effects of smoking status on immediate treatment outcomes of multidisciplinary pain rehabilitation. Pain Med. 2009 Mar;10(2):347-55. doi: 10.1111/j.1526-4637.2008.00494.x. Epub 2008 Aug 18. PMID 18721171
- See also: Mayo Pain Rehabilitation Center — http://www.mayoclinic.org/pain-rehabilitation-center-rst/research.html